CLINICAL TRIAL: NCT03136705
Title: Short-Term Effects of Nicotinamide and Lanthanum Carbonate on Phosphorus Homeostasis in Healthy Volunteers
Brief Title: Healthy Combine Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Tamara Isakova, Associate Professor Department of Medicine-Nephrology, Director of the Center for Translational Metabolism and Health, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00090161
Record Dates: First submitted 2017-03-23; First posted 2017-05-02 (Actual); Results first posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Healthy
Keywords: Phosphorus Homeostasis; FGF23; Vitamin D
MeSH Terms: interventions — Niacinamide; lanthanum carbonate; Tablets

STUDY DESIGN:
Intervention Model Description: Double blind, randomized, placebo-controlled, 2x2 factorial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Lanthanum + Nicotinamide (Active Comparator): Lanthanum Carbonate 1000mg orally three times daily with meals for 2 weeks and Nicotinamide 750mg orally twice daily for 2 weeks
  Interventions: Drug: Nicotinamide; Drug: Lanthanum Carbonate
- Lanthanum + Nicotinamide Placebo (Active Comparator): Lanthanum Carbonate 1000mg orally three times daily with meals for 2 weeks and Nicotinamide Placebo orally twice daily for 2 weeks
  Interventions: Drug: Lanthanum Carbonate; Drug: Nicotinamide Placebo
- Lanthanum Placebo + Nicotinamide (Active Comparator): Lanthanum Carbonate Placebo orally three times daily with meals for 2 weeks and Nicotinamide 750mg orally twice daily for 2 weeks
  Interventions: Drug: Nicotinamide; Drug: Lanthanum Carbonate Placebo
- Lanthanum Placebo + Nicotinamide Placebo (Placebo Comparator): Lanthanum Carbonate Placebo orally three times daily with meals for 2 weeks and Nicotinamide Placebo orally twice daily for 2 weeks
  Interventions: Drug: Lanthanum Carbonate Placebo; Drug: Nicotinamide Placebo

INTERVENTIONS:
Drug: Nicotinamide — Nicotinamide tablet
  Arms: Lanthanum + Nicotinamide; Lanthanum Placebo + Nicotinamide
Drug: Lanthanum Carbonate — Lanthanum Carbonate tablet
  Other Names: Fosrenol
  Arms: Lanthanum + Nicotinamide; Lanthanum + Nicotinamide Placebo
Drug: Lanthanum Carbonate Placebo — Sugar pill manufactured to look like Lanthanum Carbonate tablet
  Other Names: Placebo (for Lanthanum Carbonate 500mg tablet)
  Arms: Lanthanum Placebo + Nicotinamide; Lanthanum Placebo + Nicotinamide Placebo
Drug: Nicotinamide Placebo — Sugar pill manufactured to look like Nicotinamide tablet
  Other Names: Placebo (for Nicotinamide 750mg tablet)
  Arms: Lanthanum + Nicotinamide Placebo; Lanthanum Placebo + Nicotinamide Placebo

SUMMARY:
STUDY SUMMARY Title: EFFECTS OF NICOTINAMIDE AND LANTHANUM CARBONATE ON PHOSPHORUS HOMEOSTASIS Protocol Number:STU00090161 Phase: Phase 1, detailed physiologic study Methodology: double blind, randomized, placebo-controlled, 2x2 factorial Study Duration: 12-18 months (to complete the entire study protocol) Study Center: Single-center Objectives: Define short-term effects of the interventions (lanthanum carbonate and nicotinamide) on indices of phosphate handling Number of Subjects: 80 Diagnosis and Main Inclusion Criteria: Healthy volunteers Study Product(s), Dose,Route, Regimen: Nicotinamide, 750 mg by mouth twice daily, Lanthanum carbonate, Fosrenol, 1000 mg by mouth three times daily with meals Duration of administration: 2 weeks (length of time study participants are enrolled in study) Reference therapy: reference is a placebo Statistical Methodology: Repeated measures analysis using mixed linear models

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a growing public health problem that increases risks of endstage renal disease (ESRD), cardiovascular disease (CVD), fractures, and death, and it poses an enormous financial burden on the US health system. Existing therapies modestly impact outcomes. Novel strategies targeting CKD-specific mechanisms are urgently needed to improve health and reduce cost.

CKD is complicated by disordered mineral metabolism, characterized by abnormal calcium and phosphate homeostasis, calcitriol and klotho deficiency, and elevated levels of parathyroid hormone (PTH) and fibroblast growth factor 23 (FGF23). Elevated FGF23 is the earliest and most common manifestation of disordered mineral metabolism. Observational studies report independent associations between elevated phosphate and FGF23 blood levels and increased risks of ESRD, CVD and death. As potential explanatory mechanisms, phosphate excess induces arterial stiffness due to vascular calcification, and FGF23 excess contributes directly to the pathogenesis of left ventricular hypertrophy (LVH). Together, these effects promote CVD events and death.

Dietary phosphate absorption is a modifiable determinant of phosphate and FGF23 levels. Small studies of short duration suggest that phosphate binders and dietary phosphate modification in CKD can lower phosphate and FGF23 blood levels by reducing paracellular absorption of phosphate in the gut. However, animal studies demonstrate that compensatory upregulation of transcellular phosphate absorption via the sodium phosphate co-transporter, NPT2b, reduces the efficacy of these approaches. Since nicotinamide lowers plasma phosphate by reducing gut expression of NPT2b,the investigators hypothesize that use of nicotinamide combined with phosphate binders on a background of dietary phosphate moderation will most effectively reduce phosphate and FGF23 blood levels in CKD. The investigators plan to advance this approach in future randomized clinical trials.

The objective of this study is to perform a detailed physiologic study of healthy volunteers to assess the short-term effects of nicotinamide alone, lanthanum carbonate alone, or both in combination, on phosphate homeostasis. The results from healthy volunteers will provide information needed for optimal design of studies for patients with CKD.

ELIGIBILITY:
INCLUSION CRITERIA

Healthy volunteers

Age ≥ 18 years, at the time of screening

Normal renal function at screening, as defined by

* eGFR > 60
* no albuminuria
* normal urinalysis
* normotensive, defined as blood pressure <140/85mmHg
* no known history of CKD

Adequate organ and marrow function at screening as defined below:

* HCT ≥ 30%
* platelets ≥ 125,000/mm3
* total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SPGT) ≤ 2.5 X institutional upper limit
* 25-hydroxyvitamin D ≥ 10mg/dL

Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy.

Ability to understand and the willingness to sign a written informed consent.

EXCLUSION CRITERIA:

History of allergic reaction to nicotinamide, niacin (excluding flushing), and/or multivitamin preparations

Liver disease, defined as known cirrhosis by imaging or physician diagnosis.

* Documented alcohol use > 14 drinks/week
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and/or alkaline phosphatase concentrations > 2 times the upper limit of the local laboratory reference range and/or total bilirubin concentration not within institutional limits.

Creatine kinase (CK) concentrations > 2 times the upper limit of the local laboratory reference range at screening

Major hemorrhagic event within the past six months from screening requiring inpatient admission.

Blood or platelet transfusion within the past six months from screening

History of primary hyperparathyroidism

Current, clinically significant malabsorption

Anemia (screening HCT < 30%) at screening

Plasma albumin < 2.5 mg/dl at screening

25-hydroxyvitamin D <10mg/dL at screening

Inability or unwillingness to provide consent

Current or recent treatment (within the last 14 days from screening) with niacin/nicotinamide > 100 mg/day

Current or recent use of MVI containing niacin/nicotinamide > 100 mg/day

Current use of Tums (or calcium carbonate taken for indigestion) at a dose of >1000 mg daily

Current participation in another clinical trial or other interventional research

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2016-02-03 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Isakova, MD, MMSc, Principal Investigator — Northwestern University
Locations (1):
- Center for Translational Metabolism and Health (CTMH), Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Study Protocol: STU00089165 — https://irb.northwestern.edu/contact
- Available data/document: Informed Consent Form: STU00089165 — https://irb.northwestern.edu/contact

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lanthanum + Nicotinamide | Lanthanum + Nicotinamide Placebo | Lanthanum Placebo + Nicotinamide | Lanthanum Placebo + Nicotinamide Placebo
Started | 9 | 10 | 10 | 10
Completed | 9 | 10 | 10 | 9
Not Completed | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lanthanum + Nicotinamide | Lanthanum + Nicotinamide Placebo | Lanthanum Placebo + Nicotinamide | Lanthanum Placebo + Nicotinamide Placebo | Total
Number analyzed (Participants) | 9 | 10 | 10 | 10 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (15.1) | 27.1 (9.4) | 29.4 (13.4) | 26.6 (12.9) | 30.0 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 6 | 7 | 28
  Male | 2 | 2 | 4 | 3 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 5 | 9 | 7 | 6 | 27
  African American | 3 | 1 | 1 | 1 | 6
  Asian | 1 | 0 | 2 | 3 | 6
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.5 (5.2) | 23.3 (2.7) | 23.6 (3.9) | 23.2 (2.7) | 23.8 (3.7)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 109.3 (10.6) | 111.5 (12.3) | 115.8 (6.9) | 108.2 (11.6) | 111.3 (10.6)
Serum Phosphate [Mean (Standard Deviation); unit: mg/dL] | 3.4 (0.5) | 3.6 (0.4) | 3.4 (0.3) | 3.6 (0.5) | 3.5 (0.4)
Serum Creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.8 (0.2) | 0.8 (0.2) | 0.8 (0.2) | 0.8 (0.1) | 0.8 (0.2)
Urine 24 hour Phosphate total [Mean (Standard Deviation); unit: mg] | 511.8 (210.7) | 678.0 (218.8) | 799.0 (265.1) | 679.7 (244.5) | 671.1 (248.7)
Urine 24 hour Creatinine total [Mean (Standard Deviation); unit: mg] | 1114.3 (411.2) | 1505.5 (588.0) | 1646.7 (536.5) | 1489.8 (478.8) | 1447.4 (527.3)
Urine 24 hour Calcium total [Median (Inter-Quartile Range); unit: mg] | 59.6 [46.9 to 83.8] | 129.9 [118.5 to 179.9] | 175.2 [109.0 to 185.0] | 102.0 [65.0 to 123.9] | 118.5 [65.0 to 178.6]
Urine 8 hour Phosphate total [Mean (Standard Deviation); unit: mg] | 280.9 (135.0) | 377.5 (160.8) | 407.3 (184.8) | 327.6 (102.6) | 350.4 (149.8)
Urine 8 hour Creatinine total [Mean (Standard Deviation); unit: mg] | 478.5 (218.1) | 646.9 (224.3) | 687.1 (225.3) | 532.2 (116.3) | 591.8 (209.5)
Urine 8 hour Calcium total [Median (Inter-Quartile Range); unit: mg] | 50.1 [23.4 to 76.5] | 60.2 [55.8 to 87.0] | 66.4 [36.0 to 75.9] | 57.3 [42.4 to 65.6] | 59.4 [42.4 to 72.0]
Intact FGF23 [Median (Inter-Quartile Range); unit: pg/ml] | 68.0 [56.1 to 80.0] | 66.9 [41.7 to 95.5] | 54.2 [45.5 to 66.4] | 72.3 [51.6 to 100.2] | 66.2 [47.7 to 95.5]
C-terminal FG23 [Median (Inter-Quartile Range); unit: RU/ml] | 66.3 [60.9 to 84.4] | 82.1 [66.2 to 100.1] | 80.7 [54.8 to 94.1] | 90.7 [61.1 to 122.8] | 79.0 [60.9 to 100.1]

OUTCOME MEASURES:

1. Primary Outcome: Change in Intact FGF23
Description: Longitudinal change in serum intact FGF23 levels from baseline visit through completion of study.
Time Frame: Approximately 3 weeks.
Population: intention to treat
Measure: Geometric Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Lanthanum + Nicotinamide | Lanthanum + Nicotinamide Placebo | Lanthanum Placebo + Nicotinamide | Lanthanum Placebo + Nicotinamide Placebo
Number analyzed (Participants) | 9 | 10 | 10 | 9
pg/ml | 1.001 [0.978 to 1.024] | 1.006 [0.983 to 1.029] | 1.009 [0.987 to 1.032] | 1.005 [0.995 to 1.014]
Statistical Analysis 1: Comparison: Lanthanum + Nicotinamide vs Lanthanum + Nicotinamide Placebo vs Lanthanum Placebo + Nicotinamide vs Lanthanum Placebo + Nicotinamide Placebo; linear mixed model for repeated measures data; Test type: Superiority; p = 0.3738, Mixed Models Analysis; trend analysis = 1.009, 95% CI 2-sided [0.989 to 1.031]

2. Secondary Outcome: Change in Plasma Phosphorus Level
Description: Longitudinal change in plasma phosphorus levels from baseline visit through completion of study.
Time Frame: Approximately 3 weeks.
Population: intention to treat
Measure: Geometric Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Lanthanum + Nicotinamide | Lanthanum + Nicotinamide Placebo | Lanthanum Placebo + Nicotinamide | Lanthanum Placebo + Nicotinamide Placebo
Number analyzed (Participants) | 9 | 10 | 10 | 9
mg/dl | 0.0099 [-0.0407 to 0.0604] | -0.0102 [-0.0596 to 0.0392] | 0.0099 [-0.0395 to 0.0593] | 0.0004 [-0.0202 to 0.0210]
Statistical Analysis 1: Comparison: Lanthanum + Nicotinamide vs Lanthanum + Nicotinamide Placebo vs Lanthanum Placebo + Nicotinamide vs Lanthanum Placebo + Nicotinamide Placebo; linear mixed model for repeated measures data; Test type: Superiority; p = 0.854, Mixed Models Analysis; trend analysis = 0.0043, 95% CI 2-sided [-0.0414 to 0.0499]

3. Secondary Outcome: Change in 24 Hour Urinary Phosphorus Level
Description: Longitudinal change in 24 hour urinary phosphorus levels from baseline visit through completion of study.
Time Frame: Approximately 3 weeks.
Population: intention to treat
Measure: Geometric Mean (95% Confidence Interval); unit: mg
Arm/Group | Lanthanum + Nicotinamide | Lanthanum + Nicotinamide Placebo | Lanthanum Placebo + Nicotinamide | Lanthanum Placebo + Nicotinamide Placebo
Number analyzed (Participants) | 9 | 10 | 10 | 9
mg | -10.24 [-33.94 to 13.47] | -5.88 [-29.13 to 17.37] | 1.29 [-22.11 to 24.69] | -10.85 [-20.56 to -1.13]
Statistical Analysis 1: Comparison: Lanthanum + Nicotinamide vs Lanthanum + Nicotinamide Placebo vs Lanthanum Placebo + Nicotinamide vs Lanthanum Placebo + Nicotinamide Placebo; linear mixed model for repeated measures data; Test type: Superiority; p = 0.0648, Mixed Models Analysis; trend analysis = 20.38, 95% CI 2-sided [-1.26 to 42.03]

ADVERSE EVENTS:
Time Frame: Duration of the study, which with study visit windows was approximately 3 weeks
Description: Adverse event reporting did not differ from what is described under clinicaltrials.gov.
Arm/Group | Lanthanum + Nicotinamide | Lanthanum + Nicotinamide Placebo | Lanthanum Placebo + Nicotinamide | Lanthanum Placebo + Nicotinamide Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10 | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 1/10 | 0/10 | 0/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanthanum + Nicotinamide (N=9) | Lanthanum + Nicotinamide Placebo (N=10) | Lanthanum Placebo + Nicotinamide (N=10) | Lanthanum Placebo + Nicotinamide Placebo (N=9)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Hypophosphatemia, with serum phosphate level below the limit of normal, was reported in 1 participant. Study medications were held temporarily and the serum phosphate improved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT03136705/Prot_SAP_000.pdf